CLINICAL TRIAL: NCT03920878
Title: Peri- Versus Intra-operative Anti-vascular Endothelial Growth Factor Intravitreous Injections for Diabetic Macular Edema in Patients Undergoing Cataract Surgery
Brief Title: Cataract DME - Peri vs. Intraop
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study team was unable to secure sufficient funding and administrative support.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Andrew Hendrick, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00106475
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Diabetic Macular Edema; Cataract
Keywords: anti-VEGF injections; pre-existing DME; cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aflibercept injected Pre- and Post-operatively (Experimental): Pre- and Post-operative time of Aflibercept injections
  Interventions: Drug: Aflibercept injected Pre- and Post-operatively
- Aflibercept injected intraoperatively (Active Comparator): Intraoperative time of Aflibercept injection
  Interventions: Drug: Aflibercept injected intraoperatively

INTERVENTIONS:
Drug: Aflibercept injected Pre- and Post-operatively — Three injections of aflibercept before cataract surgery, and aflibercept injections after surgery within 14-21 days of the day of surgery (number of injections depends on clinical exam findings, visual acuity and retinal thickness).
  Other Names: EYELEA
  Arms: Aflibercept injected Pre- and Post-operatively
Drug: Aflibercept injected intraoperatively — Three injections of aflibercept before surgery and one injection of aflibercept during the course of the surgery by cataract surgeon.
  Other Names: EYELEA
  Arms: Aflibercept injected intraoperatively

SUMMARY:
Goals of the study are to evaluate how peri-operative versus intra-operative anti-VEGF intravitreous injections affect visual acuity (BCVA) in patients with persistent diabetic macular edema who are undergoing cataract surgery; and to evaluate how peri-operative versus intra-operative anti-VEGF intravitreous injections affect OCT CSF thickness and total number of postoperative injections in patients with diabetic macular edema who are undergoing cataract surgery.

DETAILED DESCRIPTION:
Along with age, diabetes is a major risk factor for cataract formation, which can lead to significant vision loss and disability without medical intervention. Unfortunately, diabetic patients, particularly those with diabetic macular edema (DME), experience poorer visual outcomes after undergoing cataract surgery compared to non-diabetics. Reasons for this is multifactorial but includes an increased risk in the development of post-operative cystoid macular edema, and exacerbation of baseline DME. This poses a significant challenge in managing concomitant DME and visually-significant cataracts.

Goals of the study are to evaluate how peri-operative versus intra-operative anti-VEGF intravitreous injections affect visual acuity (BCVA) in patients with persistent diabetic macular edema who are undergoing cataract surgery; and to evaluate how peri-operative versus intra-operative anti-VEGF intravitreous injections affect OCT CSF thickness and total number of postoperative injections in patients with diabetic macular edema who are undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18 with diabetes mellitus, diabetic macular edema and visually significant cataracts planning to undergo cataract surgery

Exclusion Criteria:

* Patients who have undergone panretinal photocoagulation (PRP) in prior 4 months or an ocular condition (other than cataract and DME) that might affect visual acuity during course of study.
* Patients with history of vitrectomy.
* Patients with neovascular glaucoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change in best-corrected visual acuity (BCVA) | 1 month, 3 months and 6 months after cataract surgery
  BCVA is a measurement of the best vision correction that can be achieved, such as glasses, as measured on the standard Snellen eye chart. For example, if uncorrected eyesight is 20/200, but patient can see 20/20 with glasses, the BCVA is 20/20.

SECONDARY OUTCOMES:
Change in optical coherence tomography (OCT) central subfield (CSF) thickness | 24 hours post-operatively, 1 month, 3 months and 6 months after cataract surgery
  Optical coherence tomography (OCT) is an important imaging modality in the evaluation and management of retinal diseases. Change in central subfield (CSF) thickness will be measured and recorded.
Total number of postoperative injections | 6 months after cataract surgery
  Total number of postoperative injections will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hendrick, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory Clinic, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No
No individual de-identified participant data (including data dictionaries) will be shared. Only composite results with publication will be shared.